CLINICAL TRIAL: NCT00230087
Title: Iron Depletion Therapy for Patients With Type 2 Diabetes Mellitus and Non-Alcoholic Fatty Liver Disease
Brief Title: Iron Depletion Therapy for Type 2 DM and NAFLD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Kris Kowdley MD, Virginia Mason Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DK 61728-S1 (completed)
Record Dates: First submitted 2005-09-29; First posted 2005-09-30 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Diabetes Mellitus
Keywords: diabetes; nafld; nash; phlebotomy
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus | interventions — Blood Donation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: blood donation — phlebotomy until iron depleted

SUMMARY:
The purpose of this study is to find out whether lowering the amount of iron in the body will result in less resistance to insulin and improved liver function in patients with type 2 diabetes mellitus and non-alcoholic fatty liver disease. This may result in better diabetes control and/or a decrease in the amount of liver fat.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is a common liver disease in the United States. NAFLD can lead to severe liver disease in some patients. Patients with NAFLD develop resistance to the normal action of insulin. Insulin is important for processing sugar and fat and increased resistance to insulin leads to fat in the liver. There is a correlation between the amount of iron in a person's body and the ability of insulin to work properly. Several small studies suggest that removal of iron may improve both diabetes and NAFLD by lowering insulin resistance.

The goal of this pilot study is to determine the effect of iron depletion on insulin sensitivity in patients with type 2 diabetes mellitus and non-alcoholic fatty liver disease. This study will be performed as an ancillary P&F study to the NASH CRN; all participants will be recruited from the NASH CRN Database Study. Secondary outcome measures will include the effect of iron depletion on hepatic necroinflammation, markers of oxidative stress and intrahepatic fat content. Insulin resistance will be directly measured using a two-step hyperinsulinemic euglycemic clamp procedure, before and after iron depletion by phlebotomy. Oral glucose tolerance tests will also be performed in order to evaluate the efficacy of using the indirect, but less cumbersome, HOMA model to derive values of insulin resistance in this patient cohort. This study will advance our understanding of the role of body iron stores in the pathophysiology of type 2 diabetes mellitus and non-alcoholic fatty liver disease. If iron depletion results in improved insulin sensitivity, reduced hepatic necroinflammation and/or intrahepatic fat content, a large scale, randomized, controlled trial of iron depletion in patients with type 2 diabetes mellitus and non-alcoholic fatty liver disease will be planned.

ELIGIBILITY:
Inclusion Criteria

* Histological evidence of NAFLD and enrollment in NASH CRN Database Study
* Type 2 DM treated with diet or a stable dose of non-insulin sensitizing oral hypoglycemic agents for > 3 mo.
* Hemoglobin HbA1c level ≤ 8 %
* Serum ALT levels ≥1.3 x ULN
* Between 18-65 years of age

Exclusion Criteria

* Hereditary hemochromatosis or hepatic iron overload defined as any of the following:

  * 2+ iron on hepatic iron staining
  * Hepatic Iron Index ≥ 1.9
  * C282Y homozygous or C282Y/H63D compound heterozygous HFE genotype
* Use of insulin or thiazolidinediones for the treatment of diabetes
* Use of anti-NASH drugs (thiazolidinediones, vitamin E, UDCA, SAM-e, betaine, milk thistle, gemfibrozil, anti-TNF therapies, probiotics)
* Serum ferritin <50μg/L
* Serum transferrin-iron saturation <10 %
* Hemoglobin <10 mg/L
* Hematocrit <38 %
* Voluntary blood donation or therapeutic phlebotomy within the previous twelve months (except routine lab tests)
* Pregnant or lactating women
* Prior history of coronary artery disease, myocardial infarction, exertional dyspnea or chronic chest pain at rest.
* Evidence of myocardial infarction as determined by an ECG

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2005-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Improved insulin sensitivity as determined by:(1) hyperinsulinemic euglycemic clamp method | one year
(2) HOMA model- determined by the OGTT method | one year

SECONDARY OUTCOMES:
Change in serum aminotransferase levels Change in levels of serum, plasma and urinary markers of oxidative stress | one year
Changes in intrahepatic and intraabdominal fat content as determined by CT scan | one year
Change in serum levels of proinflammatory cytokines (ie IL-6, TnF-αR2) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Kris V Kowdley, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States